CLINICAL TRIAL: NCT03023189
Title: Efficacy and Safety of Early Administration of Tranexamic Acid in Cirrhotic Patients Presenting With Acute Upper Gastrointestinal Bleeding: a Multicenter, Randomized, Double Blind, Placebo-controlled Trial (Modified by amendment1)
Brief Title: Efficacity and Safety of Tranexamic Acid in Cirrhotic Patients Presenting With Acute Upper Gastrointestinal Bleeding
Acronym: EXARHOSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P150959; 2016-002677-35 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2017-01-18 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Upper Digestive Bleeding; Cirrhosis
Keywords: Upper digestive bleeding; Haemorrhage; Cirrhosis; Antifibrinolytic; Tranexamic acid; Emergency
MeSH Terms: conditions — Fibrosis; Hemorrhage; Emergencies | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): At randomisation : loading dose of 1g of intravenous tranexamic acid for 10 min, immediately followed by an intravenous infusion of 3g of TA over 24h
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): At randomisation : loading dose of 10 mL of intravenous isotonic saline for 10 min, immediately followed by an intravenous infusion of 30 mL of isotonic saline over 24h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — At randomisation : loading dose of 1g of intravenous tranexamic acid for 10 min, immediately followed by an intravenous infusion of 3g of TA over 24h.
  Total dose : 4 g of TA
  Arms: Tranexamic acid
Drug: Placebo — At randomisation : loading dose of 10 mL of intravenous isotonic saline for 10 min, immediately followed by an intravenous infusion of 30 mL of isotonic saline over 24h Total dose : 40 mL of Placebo
  Arms: Placebo

SUMMARY:
Upper digestive bleeding. Upper gastrointestinal haemorrhage is a common cause of decompensated cirrhosis and is associated with a high mortality rate among cirrhotic patients. Its leading cause is the rupture of gastro-esophageal varices due to portal hypertension. In cirrhotic patients, the management of acute gastrointestinal haemorrhage is challenging as they often present with coagulation (or haemostasis abnormalities) abnormalities such as hyperfibrinolysis, especially when the cirrhosis is decompensated. Beyond life support measures, therapeutic modalities of upper gastrointestinal bleeding rely on both endoscopic and pharmacological interventions. Tranexamic acid (TA) is an antifibrinolytic that may help control the bleeding in this setting, as it showed an unquestionable benefit in other indications. TA has previously been studied in both upper gastrointestinal haemorrhage from any causes and in liver transplantation of cirrhotic patients. However, there is a lack of data to conclude on its effectiveness (or efficiency) in the early treatment of acute bleeding in cirrhotic patients.

Investigators hypothesize that, when given early, TA would be beneficial for cirrhotic patients presenting with acute upper gastrointestinal haemorrhage , by controlling the haemorrhage, avoiding rebleeding episodes and reducing mortality within 5 days after its administration. Moreover, TA could prevent early cirrhosis complications (such as hepatic encephalopathy, sepsis and ascites liquid infection, hepatorenal syndrome), could reduce indications to transjugular portosystemic shunt (TIPS), shorten the length of stay in intensive care unit and the length of hospitalization, and decrease late relapses and one-year mortality.

DETAILED DESCRIPTION:
Acute Upper gastrointestinal haemorrhage (UGIH) is frequent, with an estimated annual incidence of 150/100 000 in France. Its second etiology is the rupture of portal hypertension-related gastro-esophageal varices, accounting for 20 % of the patients and responsible for more than 50 % of the hospitalizations in intensive care unit (ICU) for UGIH.

In cirrhotic patients, variceal bleeding is the main cause of UGIH (over 70 %) and death (30 %), which occurs in the most severe patients (Child-Pugh score B or C and/or high MELD score, and high levels of portal hypertension).

Acute UGIH is directly responsible for 50 % of the deaths, either because it remains uncontrolled during the acute phase (within 5 days), or because of early relapses (within 6 weeks). Every episode of acute UGIH worsens the middle and long-term vital prognosis: about 60 % of the patients present with UGIH recurrence within one year and the survival rate is only 30 % 3 years after the first episode.

Moreover, acute UGIH is a triggering factor for several severe cirrhosis-specific complications (such as hepatic encephalopathy, sepsis and ascites liquid infection, hepatorenal syndrome), which themselves lead to high mortality rates. Despite the improvement of preventive, diagnostic and therapeutic strategies, UGIH remains stable in France.

The haemostasis of cirrhotic patients is often abnormal at baseline : thrombopenia, decrease of factors II, V, VII, IX, X and XI, decrease of fibrinolytic proteins, increase of factor VIII and spontaneous fibrinolysis. When compensated, the cirrhotic's haemostasis remains globally preserved, due to the balance of pro and anticoagulant alterations.

Every cause of cirrhosis decompensation, such as acute PHT-UGIH, can increase hemostatic disorders, leading to hyperfibrinolysis. This could slow down or inhibit the clotting, thus disrupting pharmacological control of acute UGIH.

TA could be efficient in acute UGIH of cirrhotic patients. It is a simple antifibrinolytic which showed clinical benefits on haemorrhage and/or mortality in several other indications (surgical, obstetrical and traumatic). It is now widely used according to recommendations.

Early administration of TA seems to be beneficial in UGIH haemorrhage. Despite theoretical efficiency, 4 recent Cochrane meta-analysis concluded to the lack of significant data (poor overall trials quality). The benefit of the use of TA in acute UGIH (and acute PHT-UGIH) remains uncertain.

At this day, TA has still not been studied in acute UGIH of cirrhotic patients, although it showed benefits on blood transfusion's requirements and on haemorrhagic complications during liver transplantation (for which cirrhosis most frequent cause).

ELIGIBILITY:
Inclusion Criteria (modified by amendment1)

* Age ≥ 18
* Patient treated by a prehospital physician-staffed SMUR team, a firefighter physician-staffed ambulance (ARBSPP), an hospital EMS or an ICU
* Acute upper digestive bleeding (< 24h) in the shape of hematemesis, described either by the physician, the patient, a relative or a member of the medical team
* Known or suspected cirrhosis (based on clinical/biological/radiographic/anamnestic data)
* Affiliated or recipient of the French social security
* Written consent (or under emergency procedures)

Exclusion Criteria (modified by amendment1)

* Known ongoing pregnancy or breastfeeding
* TA already given (if inter-hospital transfer)
* Endoscopy already performed for the current haemorrhagic episode
* Hospitalization for over 24h in an intensive care unit or a routine care unit
* Exclusive lower digestive bleeding or melena only
* Patient in cardiac arrest at the arrival of the prehospital medical team, whether recovered or not
* Patient already randomised once in EXARHOSE study
* TA Counter-indications

  * creatininemia > 500 μmol/L or documented clearance < 30 mL/min
  * documented ongoing CIVD (prior to UDB)
  * ongoing seizures
  * ongoing arterial or venous thrombosis
  * allergy
* Known participation of the patient to another therapeutic study
* Known linguistic inability of the patient to understand the study
* Patient under known guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The main outcome is a composite criterion and includes: control on acute bleeding, absence of re-bleeding episodes at day 5 and absence of death at day 5 (modified by amendment 1) | 5 days after randomisation
  Specifically, the composite criterion is defined by all the following criteria:
  * Immediate control of the hemorrhage after initial patient management using splanchnic vasoconstrictors and/or proton pump inhibitors, potentially including volume expander, transfusion and/or prescription of vasopressor amines :
  * Achievement of the transfusion target (Hb ≥ 7 g/dL) 24 hours after initial patient management and then until day 5
  * Absence of initiation or increase in vasopressor amines, until day 5
  * Absence of recourse to the transfusion of 2 or more red cells packs within 24h to maintain the transfusion target (Hb ≥ 7 g/dL)
  * Absence of persistence or evolution towards haemorrhagic shock (systolic blood pressure < 100 mmHg and/or mean arterial pressure < 60 mmHg and/or heart rate > 100 bpm)
  * Absence of re-bleeding episodes at day 5, assessed by the medical team on the bases of clinical, biological or endoscopic elements
  * Absence of death at day 5

SECONDARY OUTCOMES:
Control of the bleeding | Within 5 days after randomisation
  At least 1 criterion present :
  * Persistence of the bleeding (regardless of the volume), 2 hours after initiation of medical or endoscopic treatment
  * And/Or blood transfusion needed within 24 hours after treatment initiation (≥ 2 red cells units)
  * And/Or hemorrhagic shock installation (systolic blood pressure < 100 mmHg and/or mean arterial pressure < 60 mmHg and/or heart rate > 100 bpm)
Re-bleeding episodes | At day 6, day 28, day 42, 3 months, 6 months and 1 year after randomisation
Death | At day 6, day 28, day 42, 3 months, 6 months and 1 year after randomisation
Fluid infusion volume (in mL) | At day 6, day 28 and day 42 after randomisation
Blood transfusion volume (in mL) | At day 6, day 28 and day 42 after randomisation
Blood transfusion quantity (number of units) | At day 6, day 28 and day 42 after randomisation
Nature of blood transfusion: - Red cells units - Platelets units - Fresh frozen plasma - Fibrinogen - Other | At day 6, day 28 and day 42, after randomisation
TIPS procedure (in Child-Pugh B patients) | At day 6, day 28, day 42 after randomisation
Visceral and systemic complications | At day 6, day 28 and day 42, after randomisation (or until discharge)
  Complications, defined as:
  * Acute organ failure (using CLIF-C ACLF and CLIF-SOFA scores)
  * Hepatic encephalopathy
  * Hepatic failure
  * Hepatorenal syndrome
  * Renal failure (using grades 2 and 3 of the KDIGO classification)
  * Sepsis
  * Ascites liquid infection
Need for organ substitution - Renal replacement therapy (dialysis) - Liver replacement therapy - Mechanical ventilation | At day 6, day 28 and day 42, after randomisation (or until discharge)
Liver transplantation | At day 6, day 28, day 42, 3 months, 6 months and 1 year after randomisation
Length of stay in ICU (in days) | At day 6, day 28, day 42, 3 months, 6 months and 1 year after randomisation
Duration of hospitalization (in days) | At day 6, day 28, day 42, 3 months, 6 months and 1 year after randomisation
Number of participants with treatment-related adverse events as assessed by the ANSM notice of Exacyl® | up to 5 days
  Adverse events as assessed by the ANSM notice of Exacyl® are :
  * Allergy
  * Thrombotic events
  * Seizures
  * Acute renal failure (KDIGO grades 2 and 3)
  * Death
  * Or any other adverse event suspected to be treatment-related
  Adverse effects will be systematically searched for and collected in the electronic Case Report Form (eCRF) during the acute phase (within 5 days after randomization), as assessed by the AP-HP notification form. When present, investigators will have to send a notification to the promoter (by fax). Patients with severe adverse effects (leading to death, life-threatening condition, hospitalization and pursuit of hospitalization, incapacity or handicap, congenital malformation) will be followed until disappearance of these. Every document related to the patient during the protocol should be transmitted to the promoter. Investigators are supposed to answer every inquiry of the promoter.
Delay between the beginning of the haemorrhage and the initiation of the AT treatment | At day 1

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu HEIDET, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Jean Verdier Hospital, Bondy
  - Henri Mondor Hospital, Créteil
  - Marc Jacquet Hospital, Melun

REFERENCES:
- [Derived] Heidet M, Amathieu R, Audureau E, Augusto O, Nicolazo de Barmon V, Rialland A, Schmitz D, Pierrang F, Marty J, Chollet-Xemard C, Thirion O, Jacob L. Efficacy and tolerance of early administration of tranexamic acid in patients with cirrhosis presenting with acute upper gastrointestinal bleeding: a study protocol for a multicentre, randomised, double-blind, placebo-controlled trial (the EXARHOSE study). BMJ Open. 2018 Aug 10;8(8):e021943. doi: 10.1136/bmjopen-2018-021943. PMID 30099397
- [Derived] Heidet M, Mermet E, Vaux J, Jeremie R, Audureau E, Marty J. Simulated EMS response times until patients located in public train stations: A geospatial model to improve on-foot accessibility. Resuscitation. 2018 Oct;131:e3-e5. doi: 10.1016/j.resuscitation.2018.07.031. Epub 2018 Aug 2. No abstract available. PMID 30077741